CLINICAL TRIAL: NCT05590234
Title: Dexmedetomidine Combined With Bupivacaine for Erector Spinae Plane Block Versus Bupivacaine Alone for Postoperative Pain Control of Posterior Lumbosacral Spine Fixation Surgeries
Brief Title: Dexmedetomidine Combined With Bupivacaine for Erector Spinae Plane Block
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, engy wahsh, lecturer of clinical pharmacy, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRC-Me-2210035
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Posterior Lumbosacral Spine Fixation Surgeries
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine combined with bupivacaine group (DB group) (Active Comparator): patients received 1ug/kg dexmedetomidine plus 20 mL of bupivacaine 0.25%,
  Interventions: Drug: Dexmedetomidine injection; Drug: Bupivacaine 0.25% Injectable Solution
- bupivacaine 0.25%, (Active Comparator): patients received 20 ml of bupivacaine 0.25%
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution
- control group (S group) (Placebo Comparator): patients received 20 ml of normal saline 0.9%.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine injection — 1ug/kg dexmedetomidine plus 20 mL of bupivacaine 0.25%
  Arms: Dexmedetomidine combined with bupivacaine group (DB group)
Drug: Bupivacaine 0.25% Injectable Solution — 20 ml of bupivacaine 0.25%,
  Arms: Dexmedetomidine combined with bupivacaine group (DB group); bupivacaine 0.25%,
Drug: normal saline — 20 ml of normal saline 0.9%.
  Arms: control group (S group)

SUMMARY:
As the posterior lumbosacral spine fixation surgeries are common spine procedures done nowadays due to different causes and as this spine procedure is mostly accompanied with moderate to severe postoperative pain, so it is necessary to find an effective and efficient postoperative analgesia for patients with this surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective posterior lumbosacral spine fixation and fusion surgery due to different causes that diagnosed clinically and radiologically including MRI and Plain X ray

Exclusion Criteria:

* hypersensitivity to the drugs used in the study [local anesthetics, non-steroidal anti-inflammatory drugs, opioids and the drug under investigation (dexmedetomidine)]
* patients with any contraindication to regional anesthesia as skin infections at the site of the block
* history of bleeding disorders or receiving anticoagulant medications

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Postoperative visual analogue scale (VAS) | the first 24 hours postoperative
  The visual analog scale (VAS) is a simple and often used method for evaluating variations in pain intensity.
Amount of post operative opioid consumption for the first 24 hours | the first 24 hours postoperative
  Amount of total opioid consumption for 24 hours postoperative

SECONDARY OUTCOMES:
Postoperative visual analogue scale (VAS) | the second 24 hour postoperative
  The visual analog scale (VAS) is a simple and often used method for evaluating variations in pain intensity.
Amount of post operative opioid consumption for the second 24 hours | the second 24 hour postoperative
  Amount of total opioid consumption for the second 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Abdelmaksod Mohammed M Mousa, MD, Principal Investigator — October 6 University
Locations (1):
- October 6 university hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abu El Hassan SHA, Wahsh EA, Mousa AM, Ibrahim ARN, Mohammed EL. Comparative Study Between Dexmedetomidine with Bupivacaine and Bupivacaine Alone in Erector Spinae Plane Block for Postoperative Pain Control of Posterior Lumbosacral Spine Fixation Surgeries: A Randomized Controlled Trial. Drug Des Devel Ther. 2024 Feb 7;18:351-363. doi: 10.2147/DDDT.S444485. eCollection 2024. PMID 38344257